CLINICAL TRIAL: NCT00706043
Title: Validation of a French Translation of the Orebro Musculoskeletal Pain Screening Questionnaire (OMPSQ): A Prospective One-year Follow-up Study
Brief Title: French Validation Orebro Musculoskeletal Pain Screening Questionnaire (OMPSQ) Questionnaire
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: BA001
Record Dates: First submitted 2008-06-26; First posted 2008-06-27 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Acute Low Back Pain; Chronic Low Back Pain
Keywords: Low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Low back pain is a very common disease. Among the persons suffering of acute low back pain, about 10% are at risk of developping chronic pain. A screening questionnaire assessing this risk has been developed and validated in Swedish and English (Orebro Musculoskeletal Pain Screening Questionnaire, Linton, 2003). The aim of our study is to validate a french translation of this questionnaire. Patients suffering from acute low back pain will be asked to fill in several questionnaires at day 0, and 6 and 12 month later.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients presenting at the clinical care setting with acute low back pain
* pain lasting for less than three months
* cumulated sick leave less thant six months

Exclusion Criteria:

* unability to sufficiently read and understand French
* presence of red flags as according to the New Zealand Acute Low Back Pain Guide

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Males and females 20-55 years old suffering from acute low back pain
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-06; Primary Completion 2010-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Pain | 6 and 12 month

SECONDARY OUTCOMES:
Professional status | 6 and 12 months
functional status | 6 and 12 months